CLINICAL TRIAL: NCT01795378
Title: HLA-Haploidentical Hematopoietic Cell Transplantation and Subsequent Donor Natural Killer Cell Infusion in Refractory Acute Leukemia - A Phase 1-2a STUDY
Brief Title: Safety and Efficacy Study of Donor Natural Killer Cells Given After Haploidentical Hematopoietic Cell Transplantation
Acronym: DNKI-II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Research Institute of Bioscience & Biotechnology (Other Government)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2012-0478
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia
Keywords: acute myelogenous leukemia; acute lymphoblastic leukemia; donor natural killer cells; HLA-haploidentical hematopoietic cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: donor natural killer cell infusion — * Donor NK cells will be generated at the GCP laboratory at Asan Institute of Life Science by a team from Stem Cell Research Center, Korea Research Institute of Bioscience and Biotechnology.
  * The patients will receive donor NK cell infusion (DNKI) around on days 6 and 9 (generated from the first collection), and around on days 13 and 20 (generated from the second collection).
  * For DNKI to be given on days 6 and 9, a 3-patient cohort each will receive escalating dose of 2x10e7/kg, 5x10e7/kg, 1x10e8/kg, and 1-4 x10e8 cells.
  * The dose of DNKI to be given on days 13 and 20 will be 1-4 x10e8/kg.

SUMMARY:
The protocol treatment is to evaluate clinical effects of donor-derived natural killer cells that are given after HLA-mismatched hematopoietic cell transplantation.

DETAILED DESCRIPTION:
Those patients with acute leukemia, which is not responding to coventional chemotherapy, will be treated. The clinical effects will be evaulated in terms of safety (side effects) and anti-leukemia effect.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute leukemia, which are refractory to standard treatment. Patients should be 17 years of age or older. The performance status of the patients should be 70 or over by Karnofsky scale. Patients should not have excessive hepatic dysfunction (bilirubin less than 3.0 mg/dl, AST less than 5 times the upper normal limit).

Patients should not have excessive renal dysfunction (creatinine less than 3.0 mg/dl).

Patients should not have clinically-evident cardiac or pulmonary dysfunction. Patients and donors must sign informed consent.

Exclusion Criteria:

Patients who are pregnant or lactating are not eligible.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
occurrence and severity of side effects of donor natural killer cell infusion | 1 year

SECONDARY OUTCOMES:
anti-leukemia effect of donor natural killer cell infusion | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Lee KH, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Hwang HJ, Jung AR, Kim SH, Yun SC, Shin HJ. Reduced-intensity conditioning therapy with busulfan, fludarabine, and antithymocyte globulin for HLA-haploidentical hematopoietic cell transplantation in acute leukemia and myelodysplastic syndrome. Blood. 2011 Sep 1;118(9):2609-17. doi: 10.1182/blood-2011-02-339838. Epub 2011 Jun 28. PMID 21715313
- [Background] Yoon SR, Lee YS, Yang SH, Ahn KH, Lee JH, Lee JH, Kim DY, Kang YA, Jeon M, Seol M, Ryu SG, Chung JW, Choi I, Lee KH. Generation of donor natural killer cells from CD34(+) progenitor cells and subsequent infusion after HLA-mismatched allogeneic hematopoietic cell transplantation: a feasibility study. Bone Marrow Transplant. 2010 Jun;45(6):1038-46. doi: 10.1038/bmt.2009.304. Epub 2009 Nov 2. PMID 19881555